CLINICAL TRIAL: NCT01207752
Title: Evaluation of the Efficacy of an Ocular Emulsion on the Signs and Symptoms of Meibomian Gland Dysfunction
Brief Title: The Efficacy of an Ocular Emulsion in Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jerry Paugh, Professor Emeritus, Southern California College of Optometry at Marshall B. Ketchum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCCO 10-6
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Meibomian Gland Dysfunction
Keywords: dry eye, MGD, tear film break up time
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes | interventions — Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Balance (Experimental): Artificial tear emulsion
  Interventions: Drug: Systane Balance
- Optive Lubricant Eye Drops (Active Comparator): Artificial tear
  Interventions: Drug: Optive Lubricant Eye Drops

INTERVENTIONS:
Drug: Systane Balance — Artificial tear emulsion drop
  Arms: Systane Balance
Drug: Optive Lubricant Eye Drops — Artificial tear eye drop
  Other Names: Refresh Optive
  Arms: Optive Lubricant Eye Drops

SUMMARY:
The aim of this study will be to determine the efficacy of this novel, lipid-containing artificial tear on the signs and symptoms of meibomian gland disease.

DETAILED DESCRIPTION:
This investigation will involve approximately 90 MGD subjects, randomly assigned to either the Systane Balance treatment group or a control group using Optive™ Lubricant Eyedrops (Allergan), a low-viscosity artificial tear. Both arms will dose the drops four times per day and the treatment trial will be conducted for 6 months. The age range will be 18 years and older, with no upper age limit. Standard diagnostic tests for dry eye, as recommended by the NEI-Industry Workshop report,8 but with updated criteria in some instances, will be used to define clinical dry eye of the MGD sub-type. The three major tests will be: symptoms using a validated questionnaire (Schein), evidence of ocular surface damage, and demonstration of tear instability. The subjects will be enrolled if they consent and are confirmed as MGD subjects using the established clinical criteria used at SCCO of gland dropout Grade 1 per lower eyelid using meiboscopy,6, 9 or secretion quality Grade 1 in any of the three sectors (temporal, central, nasal) upon gland expression9, 10 using the recently developed Korb device.11 The principal outcome measure will be the tear film breakup time (TBUT), in seconds, at two hours post drop instillation. The two-hour TBUT value will be used to compare the control and test formulation at baseline and visits 3, 5 and 7. TBUT will be measured using 2.0 l of 1.0% NaFl. Exploratory outcome measures will include TBUT (seconds; change over time), corneal staining (change over time; 0 - 20 scale), symptoms (Schein and MGD-specific preliminary questionnaire score), drop comfort, Surface Regularity Index (a measure of surface disruption), lipid layer grade (1 - 5 Yokoi scale), meibum excreta quality, gland drop out and lid margin appearance all monitored as the change over time from baseline. Treatment comparisons will be made at each timepoint

ELIGIBILITY:
Inclusion Criteria:

* Schein symptom score (all 6 questions) of greater than 5,
* evidence of MGD changes in both eyes (i.e.,
* lower eyelid secretion quality score greater than 1.0 (0 - 3 scale) OR gland dropout score greater than 1.0 (i.e., greater than 25% of entire lower eyelid) as demonstrated by meiboscopy, and corneal staining of grade 4.0 or greater (0 - 20 scale).

Exclusion Criteria:

* contact lens wear, use of topical ocular medication other than artificial tears (use of Restasis is specifically excluded),
* unstable systemic medication use (i.e., anti-histamines, steroids, etc.), recent (within 6 months of study start) ocular trauma or surgery,
* diabetes, aqueous deficient dry eye (defined as a Schirmer I value (without anesthetic) of < 5 mm of wetting in 5 minutes in either eye), and use of punctal plugs.

-Subjects taking omega 3 fatty acid supplements for dry eye can be included so long as their intake is stable for the prior six months and they meet the inclusion criteria above. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Paugh, OD, PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Eye Care Center, Fullerton, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Systane Balance | Optive Lubricant Eye Drops
Started | 35 | 34
Completed | 33 | 27
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Balance | Optive Lubricant Eye Drops | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 34 | 69
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (17.7) | 54.7 (17.5) | 52.7 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 24 | 54
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Breakup Time
Description: time in seconds to observer a dark spot in the tear film
Time Frame: Measured 2 hours after in-office administration of a single drop of test solution
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Systane Balance | Optive Lubricant Eye Drops
Number analyzed (Participants) | 32 | 28
seconds | 4.65 (1.73) | 4.42 (1.14)
Statistical Analysis 1: Comparison: Systane Balance vs Optive Lubricant Eye Drops; Test type: Superiority or Other; p = 0.550, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Systane Balance | Optive Lubricant Eye Drops
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other